CLINICAL TRIAL: NCT05040451
Title: The EXERCISE FMR Trial: An Initial Evaluation of the Carillon Mitral Contour System for Treatment of Exercise Induced Functional Mitral Regurgitation
Brief Title: Carillon Mitral Contour System for Treatment of Exercise Induced Functional Mitral Regurgitation
Acronym: EXERCISE FMR
Status: Withdrawn | Type: Observational
Why Stopped: Lack patients and site resources for the proposed population
Sponsor: Cardiac Dimensions Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CVP-3500-01
Record Dates: First submitted 2021-05-13; First posted 2021-09-10 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Carillon Mitral Contour System — The Carillon Mitral Contour System (XE2) consists of the following components:
  * An implant intended for permanent placement in the coronary sinus (CS)/great cardiac vein (GCV)
  * A delivery system which consists of a custom 9F delivery catheter and a handle assembly.

SUMMARY:
Evaluate the hemodynamic and anatomical effect of the commercially available CMCS system within its current indication on a subset of patients with exercise induced mitral regurgitation. This will be primarily evaluated by standard of care exercise testing and echocardiography. The purpose is to evaluate HFrEF CHF patients that may have mild to moderate-severe MR at rest but aggravated upon activity.

DETAILED DESCRIPTION:
The EXERCISE FMR trial is a prospective, multi-center clinical trial.

The centers will utilize pre-screening of existing medical records to identify potentially eligible subjects. Once informed consent has been obtained, the subject will undergo standard of care assessments which include: Transthoracic echocardiography, transesophageal echocardiography (if necessary), and functional assessments (NYHA and KCCQ Quality of Life Questionnaire). Following final eligibility determination, eligible subjects will under the index procedure to implant the commercially available Carillon device (includes coronary sinus venogram) according to the Instructions for Use. Subject will be discharged following after standard of care discharge assessments are completed.

Implanted subjects will have follow-up assessments performed at 1 month, 6 months, and 12 months post index procedure. Most assessments performed as part of follow-up are intended to be standard of care at each institution. The only elements that may fall outside of standard of care would be the non-invasive assessments of TTE, 6-minute walk test and the questionnaire. Further, follow-up at 1 and 6 months may also not be common site practice.

ELIGIBILITY:
Inclusion Criteria:

* Mild-moderate-to-severe secondary MR (as assessed by qualitative, semi-quantitative and/or quantitative echocardiographic assessment (Zoghbi, JASE 2017)) in the setting of all of the following (a-d, below):

  1. Symptomatic functional (secondary mitral regurgitation defined as both: 1+ (mild) 2+ (Moderate), or 3+ (Moderate/Severe)
  2. Exacerbation of MR with exercise by at least one grade or 10 mm2 EROA
  3. Left Ventricular Ejection Fraction ≤50% by Simpson's biplane technique
  4. LVEDD >5.5 cm
* New York Heart Association (NYHA) Class II, III or ambulatory IV heart failure
* Stable heart failure medication regimen for at least 30 days prior to index procedure
* Patient deemed appropriate candidate for transcatheter mitral valve repair by the local multidisciplinary heart team
* Subject meets anatomic screening criteria as determined by angiographic screening at the time of the index procedure to ensure that implant can be sized and placed in accordance with the Instructions for Use
* Female subjects of child-bearing potential must have a negative serum βHCG test
* Age ≥ 18 years old
* The subject has read the informed consent, agrees to comply with the requirements, and has signed the informed consent to participate in the study

Exclusion Criteria:

* Hospitalization in past three (3) months due to myocardial infarction, coronary artery bypass graft surgery, and/or unstable angina
* Evidence of transient ischemic attack or stroke within three (3) months prior to intervention
* Percutaneous coronary intervention in the last 30 days
* Subjects expected to require any cardiac surgery, including surgery for coronary artery disease or for pulmonic, aortic, or tricuspid valve disease within one (1) year
* Subjects expected to require any percutaneous coronary intervention within 30 days of the index procedure.
* Pre-existing device (e.g., pacing lead) in coronary sinus (CS) / great cardiac vein (GCV), or anticipated need for cardiac resynchronization therapy (CRT) within twelve (12) months
* Presence of a coronary artery stent under the CS / GCV in the implant target zone
* Presence of left atrial appendage (LAA) clot.
* Presence of primary renal dysfunction or significantly compromised renal function as reflected by a serum creatinine > 2.2 mg/dL (194.5 μmol/L) OR estimated Glomerular Filtration Rate (eGFR) < 30 ml/min
* Poorly controlled atrial fibrillation or flutter, with poor ventricular rate control (> 100 bpm resting HR), or other poorly controlled symptomatic brady- or tachy-arrhythmias
* Uncontrolled hypertension (BP > 180 mmHg systolic and/or >105 mmHg diastolic) or hypotension (BP < 90 mmHg systolic) at baseline
* Presence of severe mitral annular calcification
* Prior mitral valve surgery
* Presence of a mechanical mitral heart valve, mitral bio-prosthetic valve or mitral annuloplasty ring
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Active endocarditis
* Severe aortic stenosis (aortic valve area <1.0 cm2) or severe aortic regurgitation
* Infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, sarcoidosis)
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than functional mitral regurgitation
* Subjects with echocardiographic documentation of non-compaction cardiomyopathy with associated hypercontractility of the cardiac structures supporting the mitral annulus
* Hemodynamic instability requiring inotropic support or mechanical heart circulatory support
* Active infections requiring current antibiotic therapy
* Severe right ventricular failure or severe tricuspid regurgitation
* History of bleeding diathesis or coagulopathy, or subject who refuses blood transfusions
* Significant organic mitral valve pathology (e.g., moderate or severe myxomatous degeneration, with or without mitral leaflet prolapse, rheumatic disease, full or partial chordal rupture)
* Allergy to contrast dye that cannot be pre-medicated
* Pregnant or planning pregnancy within next 12 months.
* Chronic severe pathology limiting survival to less than 12-months in the judgement of the investigator
* Anticipated need of left ventricular assist device within twelve (12) months
* Currently participating or has participated in another investigational study where the study primary endpoint was not reached at the time of screening
* Patient requires emergent/emergency treatment for mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consent up to 150 subjects suffering from heart failure and presenting with functional mitral regurgitation in order to implant 30 subjects, plus up to 3 "roll-in" subjects per site
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in MR Volume | 6 Months
  Change in mitral regurgitant volume (mL) associated with the Carillon device from rest and exercise at 6 months post-implant, as compared to baseline

SECONDARY OUTCOMES:
Change of MR Severity: Quantitative MR Variables | 1, 6 & 12 Months
  MR severity as assessed by echocardiography in hospital, 1 month, 6 months and 12 months, in accordance with American Society of Echocardiography guidelines, compared to baseline. Quantitative MR variables to be assessed include regurgitant volume (mL), regurgitant fraction (%) and effective regurgitant orifice area (cm2, EROA) by Proximal Isovelocity Surface Area (PISA).
Change of MR severity: Semi-Quantitative Parameter (1) | 1, 6 & 12 Months
  Change in vena contract width. MR severity as assessed by echocardiography in hospital, 1 month, 6 months and 12 months, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change of MR severity: Semi-Quantitative Parameter (2) | 1, 6 & 12 Months
  Change in MV EVmax. MR severity as assessed by echocardiography in hospital, 1 month, 6 months and 12 months, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change of MR severity: Semi-Quantitative Parameter (3) | 1, 6 & 12 Months
  Change in pulmonary vein flow. MR severity as assessed by echocardiography in hospital, 1 month, 6 months and 12 months, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change in Left Atrial Area | 1, 6 & 12 Months
  Change in Left Atrial Area as assessed by echocardiography at 1, 6 and 12 months over baseline
Change in Left Atrial Diameter | 1, 6 & 12 Months
  Change in Left Atrial Diameter as assessed by echocardiography at 1, 6 and 12 months over baseline
Change in Left Atrial Volume Index | 1, 6 & 12 Months
  Change in Left Atrial Volume as assessed by echocardiography Index at 1, 6 and 12 months over baseline
Change in Left Ventricular End Systolic Volume (LVESV) | 1, 6 & 12 Months
  Change in Left Ventricular End Systolic Volume (LVESV) as assessed by echocardiography at 1, 6 and 12 months over baseline
Change in Pulmonary Artery Systolic Pressure | 1, 6 & 12 Months
  Change in Pulmonary Artery Systolic Pressure as assessed by echocardiography at 1, 6 and 12 months over baseline
Change in Quality-of-Life Overall Score | 1, 6 & 12 Months
  Change in Quality of Life (QoL) score, as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) at 1, 6 and 12 months over baseline
Change in NYHA | 1, 6 & 12 Months
  Change in New York Heart Association (NYHA) Functional Classification at 1, 6 and 12 months over baseline
Rate of Heart Failure Hospitalizations | 1, 6 & 12 Months
  Rate of hospitalization for heart failure at 1, 6 and 12 months
Rate of Major Cardiovascular Events | 1, 6 & 12 Months
  Rate of stroke, myocardial infarction, cardiovascular and all-cause mortality at 1, 6 and 12 months
Rate of Other Mitral Valve Interventions | 1, 6 & 12 Months
  Number of participants in need of mitral valve intervention or surgery at 1, 6 and 12 months

IPD SHARING:
Plan to Share IPD: No
No plans for sharing